CLINICAL TRIAL: NCT01521338
Title: G551D Observational Study (GOAL)-Expanded to Additional Genotypes and Extended for Long Term Follow up (GOAL-e2)
Brief Title: G551D Observational Study- Expanded to Additional Genotypes and Extended for Long Therm Follow up (GOAL-e2)
Acronym: GOAL- e2
Status: Completed | Type: Observational
Sponsor: Steven M Rowe (Other)
Responsible Party: Sponsor-Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: F11120200
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; G551D; G551D Mutation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Sputum, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this research study is to collect blood and urine samples from people who have either the R117H type of CF or the non-G551D gating type of CF to be kept for future research.We will also use some of the collected blood to measure the number of neutrophils.

DETAILED DESCRIPTION:
* Blood Collection: Blood will be collected to be kept for research in the future and to measure the number of blood cells called neutrophils. A small needle will be used to collect blood from a vein in your arm. About 7-9 teaspoons of blood would be collected.
* Sweat Collection: Your sweat will be collected with a special sweat collection machine to test the amount of salt in your sweat.
* Spirometry: You will be asked to take a test that measures how well your lungs are working. You will be asked to take a deep breath and then blow into a mouthpiece as hard as possible and for as long as possible. This is the same test that is done when you come to clinic.
* Urine Collection: Urine will also be collected to be kept for research in the future. You will be asked to pee in a cup.
* Medical Information: We are asking you to share your medical information with study researchers. Your medical information will not contain any of your personal identification information, like your name and address.

Optional:

• Induced Sputum Collection: If you say "yes" to collecting a sputum sample, you will be asked to breathe in a salt water solution to help you cough out sputum. If you cannot breathe in the salt water solution to cough out sputum for the last study visit, you will be asked to cough mucus into a cup

ELIGIBILITY:
Inclusion Criteria for Core Study:

1. Male or female ≥ 6 years of age at Visit 1. :
2. Must have a clinical diagnosis of cystic fibrosis and the following CFTR mutations:

   1. For Cohort 1 (Closed to enrollment June 30, 2012):

      G551D on at least 1 allele Any known or unknown mutations allowed on second allele.
   2. For Cohort 2:

      R117H on at least 1 allele Any known or unknown mutation on the second allele except G551D
   3. For Cohort 3:

   A Non-G551D gating mutation on one allele: (G178R, S549N, S549R, G551S,G970R, G1244E, S1251N, S1255P, G1349D) Any known or unknown mutation on the second allele except G551D OR R117H
3. Enrolled in the Cystic Fibrosis Foundation Patient Registry (with the exception of Canadian sites). (Patients may enroll in the Registry at Visit 1 if not previously enrolled.)
4. Clinically stable with no significant changes in health status within the 14 days prior to Visit 1.
5. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.

Exclusion Criteria for Core Study

1. Participation in the VX-770-105, VX-770-106, VX-770-108, VX-770-110, VX-770-111, VX-770-112, or VX-770-113 study, VX-770 Extended Access Program or use of ivacaftor within 6 months prior to Visit 1.
2. Any upper or lower respiratory symptoms requiring treatment with oral, inhaled or IV antibiotics within the 2 weeks prior to Visit 1.
3. History of solid organ transplantation.
4. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cystic Fibrosis and the G551D, R117H and non-G551D gating Mutations ages 6 years old and older
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint for the Core Study | Change in FEV1% predicted between Visit 1 and Visit 5
  Change in FEV1% predicted between Visit 1 and visit 5

SECONDARY OUTCOMES:
Change in sweat chloride between Visit 1 and Visit 5. | VISIT 1 AND VISIT 5
  Change in sweat chloride between Visit 1 and Visit 5.
Change in body weight between Visit 1 and Visit 5. | VISIT 1 AND VISIT 5
  Change in body weight between Visit 1 and Visit 5.

OTHER OUTCOMES:
ASSOCIATION BETWEEN PRIMARY AND SECONDARY ENDPOINTS | 1 YEAR
  The core and sub-studies will be linked so that associations between primary and secondary endpoints from each sub-study and clinical parameters (e.g., spirometry, weight, and sweat chloride) collected as part of the Core Study may be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Rowe, MD, Principal Investigator — University of Alabama at Birmingham
Locations (36):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - The Children's Hospital Colarado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children Indiana University Medical Center, Indianapolis, Indiana
  - Indianapolis University, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - The Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Grand Rapids CF Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital--University of Missouri at Kansas City, Kansas City, Missouri
  - Dartmouth Hitchcock Clinic-Lebanon, Lebanon, New Hampshire
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nation Wide Childrens Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC- University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern/Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Intermountain Cystic Fibrosis Center University of Utah Health Sciences Center, Salt Lake City, Utah
  - West Virginia University CF Medical Center, Morgantown, West Virginia
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Donaldson SH, Laube BL, Corcoran TE, Bhambhvani P, Zeman K, Ceppe A, Zeitlin PL, Mogayzel PJ Jr, Boyle M, Locke LW, Myerburg MM, Pilewski JM, Flanagan B, Rowe SM, Bennett WD. Effect of ivacaftor on mucociliary clearance and clinical outcomes in cystic fibrosis patients with G551D-CFTR. JCI Insight. 2018 Dec 20;3(24):e122695. doi: 10.1172/jci.insight.122695. PMID 30568035
- [Derived] van de Peppel IP, Doktorova M, Berkers G, de Jonge HR, Houwen RHJ, Verkade HJ, Jonker JW, Bodewes FAJA. IVACAFTOR restores FGF19 regulated bile acid homeostasis in cystic fibrosis patients with an S1251N or a G551D gating mutation. J Cyst Fibros. 2019 Mar;18(2):286-293. doi: 10.1016/j.jcf.2018.09.001. Epub 2018 Sep 29. PMID 30279125